CLINICAL TRIAL: NCT05389306
Title: Combining MRI Scanning and Contrast-Enhanced Ultrasonography to Diagnose Small Cervical Lymph Node Metastases in Patients With Nasopharyngeal Carcinoma
Brief Title: Combining MRI and CEUS to Diagnose Small Cervical Lymph Node Metastases in NPC Patients
Acronym: NPC-LN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-FXY-041-FLK
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Lymph Node; Diagnosis; Contrast-Enhanced Ultrasonography; Magnetic Resonance Imaging; Sonazoid
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Scanning and CEUS for detection of small cervical lymph node metastases. (Experimental): All patients enrolled will undergo an MRI Scanning and CEUS to evaluate their cervical lymph nodes. Ultrasound-guided lymph node aspiration and pathologic examination will be performed subsequently to obtain definitive diagnosis of the lymph nodes. The pathologic results of the lymph nodes will be adopted as gold standard to evaluate the diagnostic performance of MRI Scanning, CEUS, and the combined diagnostic criteria.
  Interventions: Diagnostic Test: MRI Scanning; Diagnostic Test: Contrast-Enhanced Ultrasonography; Diagnostic Test: Ultrasound-guided Lymph Node Aspiration

INTERVENTIONS:
Diagnostic Test: MRI Scanning — MRI scanning will be performed with a 3.0-T magnetic resonance imaging system with a head and neck-combined coil employing spin-echo technique. The range of the MRI scanning will be from the suprasellar cistern to the inferior margin of the sternal end of the clavicle. The section thicknesses for the axial plane, the sagittal plane and the coronal plane will be 5 mm, 3 mm and 2 mm, respectively. The intersection gaps will be 1 mm. Before the intravenous injection of the MRI contrast agents, T1 weighted images, T2 weighted images and diffusion weighted images will be obtained in the axial planes, while only T1 weighted images will be obtained in the sagittal and coronal planes. After the intravenous injection of the MRI contrast agents, T1-weighted axial sequence, T1-weighted sagittal sequences and T1-weighted fat-suppressed coronal sequence will be performed.
Diagnostic Test: Contrast-Enhanced Ultrasonography — A sonographer equipped with a 6-15 MHz linear array probe will be adopted for contrast-enhanced ultrasonography examination. Conventional high-frequency ultrasonography will be performed firstly before the intravenous injection of the ultrasound contrast agents. Then the ultrasound contrast agents will be injected intravenously, and contrast-enhanced ultrasonography examination will be performed. The mechanical index of contrast-enhanced ultrasonography examination will be 0.23. The wash-in and wash-out process within the lymph node will be dynamically observed during the arterial phase. During the Kupffer-phase, the degree of enhancement will also be observed.
Diagnostic Test: Ultrasound-guided Lymph Node Aspiration — After the conventional high-frequency ultrasonography and contrast-enhanced ultrasonography examination was finished, ultrasound-guided aspiration of the target lymph node will be performed. The lymph node tissue obtained from ultrasound-guided lymph node aspiration will be subjected to pathologic evaluation. And the diagnostic performance of MRI and contrast-enhanced ultrasonography will be evaluated using the pathologic diagnosis of the lymph node as the gold standard.

SUMMARY:
This is a single-center diagnostic accuracy study, with the purpose to define the criteria to diagnose small cervical lymph node metastases in patients with nasopharyngeal carcinoma by combining MRI scanning and contrast-enhanced ultrasonography and evaluate the diagnostic performance of the criteria.

DETAILED DESCRIPTION:
For newly diagnosed and histologically confirmed nasopharyngeal carcinoma patients staged as T1-4, N0-1/N3, M0 (AJCC 8th), if no metastatic lymph nodes were found on MRI according to the current diagnostic criteria, but there were small lymph nodes with a minimal axial diameter ≥ 5 mm (6 mm for lymph node in level IIA) on at least one side of the patient's neck, they will be eligible for this study. The MRI image of the small lymph nodes will be evaluated in details by experienced radiologists. Contrast-enhanced ultrasonography with specific ultrasound contrast agents (Sonazoid) and ultrasound-guided lymph node aspiration will be performed. Subsequently, the lymph node tissue obtained from ultrasound-guided lymph node aspiration will be subjected to pathologic evaluation. Using the pathologic diagnosis of the lymph node as the gold standard, diagnostic performance of MRI and contrast-enhanced ultrasonography will be evaluated. Resonable criteria to diagnose small cervical lymph node metastases by combining MRI scanning and contrast-enhanced ultrasonography will be explored. And the diagnostic performance of the criteria will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status ≤1;
2. Patients with histologically confirmed nasopharyngeal carcinoma;
3. Tumor staged as T1-4, N0-1/N3, M0 (AJCC 8th);
4. On at least one side of the patient's neck, no metastatic lymph nodes were found on MRI according to the current diagnostic criteria, but there were small lymph nodes with a minimal axial diameter ≥ 5 mm (6 mm for lymph node in level IIA);
5. Patients must be informed of the investigational nature of this study and give written informed consent. And they should be willing and able to comply with the requirements of examination, treatment, follow-up and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. History of other malignant tumors, except for adequately treated basal cell carcinoma, squamous cell carcinoma and cervical carcinoma in situ;
2. Previous radiotherapy, except radiotherapy for non-melanoma skin cancer outside the neck or nasopharyngeal regions;
3. Patients with coexistent head and neck squamous cell carcinoma besides nasopharyngeal carcinoma;
4. Patients with coexistent acute inflammation or infection (including infection within the area for aspiration);
5. Previous surgery or trauma within the neck or nasopharyngeal regions;
6. Not suitable for aspiration due to abnormal coagulation function;
7. All the candidate small lymph nodes with a minimal axial diameter ≥ 5 mm (6 mm for lymph node in level IIA) were not suitable for aspiration owing to high risk of severe complications after the aspiration；
8. Contraindications for the examination specified in the research schedule due to claustrophobia, the presence of metal implants or pacemaker, and allergic hypersensitivity to ultrasound contrast agents or MRI contrast agents;
9. Other situation assessed by the investigators that may compromise the safety or compliance of patients, such as serious disease requiring timely treatment (including mental illness), severe laboratory abnormalities, or family-social risk factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined Diagnostic Criteria to Diagnose Small Cervical Lymph Node Metastases | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.
  The criteria to diagnose small cervical lymph node metastases in patients with nasopharyngeal carcinoma by combining MRI scanning and contrast-enhanced ultrasonography with specific ultrasound contrast agents (Sonazoid).
Sensitivity and Specificity of the Combined Diagnostic Criteria | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.

SECONDARY OUTCOMES:
Receiver Operating Characteristic Curve and Optimal Cut-off Value of Each Characteristics of Small Lymph Nodes in MRI Scanning and CEUS Examination | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.
  The receiver operating characteristic curve of each characteristics of small lymph nodes in MRI scanning and CEUS examination will be plotted. The area under the curve will be calculated. And the optimal cut-off value of each characteristics will be determined based on the receiver operating characteristic curve.
Diagnostic Performance of Each Characteristics of Small Lymph Nodes in MRI Scanning and CEUS Examination Based on the Optimal Cut-off Value | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.
  The diagnostic performance of each characteristics of small lymph nodes in MRI scanning and CEUS examination will be evaluated with sensitivity, specificity, Youden index, accuracy, positive predictive value, negative predictive value, positive likelihood ratio, and negative likelihood ratio.
Inter-operator Agreement of Each Characteristics of Small Lymph Nodes in MRI Scanning and CEUS Examination | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.
  The inter-operator agreement of qualitative characteristics of small lymph nodes in MRI scanning and CEUS examination will be evaluated with Cohen's kappa coefficient. The inter-operator agreement of quantitative characteristics of small lymph nodes in MRI scanning and CEUS examination will be evaluated with Bland-Altman analysis and paired t-test.
Diagnostic Performance of the Combined Diagnostic Criteria | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.
  The diagnostic performance of the combined diagnostic criteria will be evaluated with area under the receiver operating characteristic curve, Youden index, accuracy, positive predictive value, negative predictive value, positive likelihood ratio, and negative likelihood ratio.
Inter-operator Agreement of the Combined Diagnostic Criteria | The pathologic results of the lymph nodes are expected to be obtained within one week after the MRI scanning, CEUS examination, and ultrasound-guided lymph node aspiration.
  The inter-operator agreement of the combined diagnostic criteria will be evaluated with Cohen's kappa coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No